CLINICAL TRIAL: NCT03320473
Title: A Prospective Study of Small Aperture Intraocular Lens (IOL) Implantation in KAMRA Inlay Patients After Inlay Removal
Brief Title: IOL Implantation After KAMRA Inlay Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AcuFocus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC-8 302 KAMR
Record Dates: First submitted 2017-10-22; First posted 2017-10-25 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cataract; Presbyopia
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IC-8 IOL (Experimental): IC-8 IOL implantation after removal of KAMRA ACI 7000 PDT inlay
  Interventions: Device: IC-8 IOL

INTERVENTIONS:
Device: IC-8 IOL — The AcuFocus IC-8 intraocular lens (IC-8 IOL) is a one-piece hydrophobic acrylic posterior chamber IOL into which a circular mask with a small 1.36 mm central aperture has been embedded. The IOL mask works by extending the depth of focus and its design is based on the KAMRA corneal inlay, which operates under the principle of small aperture optics.

SUMMARY:
A. The primary purpose of the study is to evaluate outcomes of aphakic eyes implanted with the IC-8 IOL following cataract removal in prior inlay patients after KAMRA inlay removal.

B. The secondary purpose of the study is to determine whether there are any changes in biometry measurements before and after the inlay removal and how the changes affect the calculated IOL power.

DETAILED DESCRIPTION:
This will be a prospective study in which no more than 20 subjects will be implanted with IC-8 IOL following the removal of the KAMRA inlay. The refractive target of the IC-8 eye will be -0.75 D MRSE.

Subjects will be screened for eligibility and consented before enrolled. Following enrollment, the inlay will be removed, and the eye will be monitored for corneal and refractive stability before the implantation of the IC-8 IOL. Corneal stability is defined as keratometry readings in each meridian within ± 0.50 D, and/or the stability of the corneal topography as determined by the principal investigator, over two consecutive visits at least two weeks apart. Refractive stability is defined as manifest refractive sphere and cylinder measurements that are each within ± 0.50 D over two consecutive visits at least two weeks apart, or based on investigator judgment. When corneal and refractive stability are achieved, the IC-8 IOL will be implanted following cataract extraction by phacoemulsification.

ELIGIBILITY:
Inclusion Criteria:

i. Subjects must sign and be given a copy of the informed consent form. ii. Subjects with BCDVA of 20/40 or worse, or significant visual symptoms/complaints as a result of cataract in the study eye.

iii. Subjects must be > 45 years of age at the time of screening. iv. Subjects must be willing and able to return for scheduled follow up examinations for 12 months after surgery.

v. Subjects who underwent uneventful KAMRA inlay implantation and who currently still have the inlay in the eye.

vi. Potential visual acuity following cataract removal and IOL implantation projected to be 0.8 or better (Snellen 20/25) as determined by diagnostic testing or investigator's medical judgment.

Exclusion Criteria:

i. Patients who had any type of intraocular surgery or refractive surgery (with the exception of KAMRA inlay implantation).

ii. Requiring an intraocular lens outside the available power range of +15.5 to +27.5 diopters.

iii. Pharmacologically dilated pupil size less than 6 mm or the presence of any pupil abnormalities (aniridia, non-reactive, fixed, or abnormally shaped pupils) or marked microphthalmos.

iv. Preoperative corneal astigmatism > 1.5 diopters (as determined by corneal topography or keratometry in either eye) or irregular corneal astigmatism.

v. Corneal abnormalities such as stromal, epithelial or endothelial dystrophies, or diagnosed degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that are predicted to cause visual acuity losses to a level of 0.8 or worse during the study.

vi. Active or recurrent anterior segment pathology (chronic uveitis, iritis, iridocyclitis, rubeosis iridis, etc.).

vii. Glaucoma suspect, uncontrolled ocular hypertension, or history of glaucomatous changes in the retina or visual field.

viii. Subjects with uncontrolled systemic disease. ix. Subjects with previous retinal pathology in either eye.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
BCDVA | 3 months
  Mean monocular best-corrected distance visual acuity at three months is at least 0.3 logMAR

SECONDARY OUTCOMES:
UCNVA | 3 months
  b.1. Mean monocular uncorrected near visual acuity (UCNVA) at 40 cm at 3 months is at least 0.3 logMAR.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Tarantino, OD, Study Director
Locations (1):
- Asian Eye Institute, Makati City, Philippines

IPD SHARING:
Plan to Share IPD: Undecided